CLINICAL TRIAL: NCT06598124
Title: Assessing the Effects of Low Lactose Milk Containing GOS (Galactooligosaccharides) on Digestive Response in Healthy Chinese Adults
Brief Title: Effects of Low Lactose Milk Containing GOS on Digestive Response in Healthy Chinese Adults
Acronym: MilkRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2314NR
Record Dates: First submitted 2024-08-15; First posted 2024-09-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Lactose; GOS; Digestive response; Gut comfort

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, 2x2 cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Other): Visit 1: Comparator Product; Visit 2: Investigational Product
  Interventions: Other: Investigational Product (IP); Other: Comparator Product (CP)
- Arm 2 (Other): Visit 1: Investigational Product; Visit 2: Comparator Product
  Interventions: Other: Investigational Product (IP); Other: Comparator Product (CP)

INTERVENTIONS:
Other: Investigational Product (IP) — 1 single dose of IP consisting in 400 mL of milk with low lactose content and GOS.
Other: Comparator Product (CP) — 1 single dose of CP consisting in 400 mL of milk with lactose

SUMMARY:
We are aiming to assess the effects of low lactose milk containing galactooligosaccharides (GOS) on digestive response in healthy Chinese adults in comparison with a matching milk containing lactose.

DETAILED DESCRIPTION:
This is planned to be single-center, double-blind, randomized, 2x2 cross-over study.

24 healthy participants of Chinese ethnicity are planned to be enrolled. Participants will be invited to three visit days at the research site: a screening visit and two test days, 3 to 28 days apart.

During the test days, participants will be requested, after overnight fasting, to consume either the investigational product (IP), a skimmed milk powder with low lactose content and GOS, or the comparator product (CP) a matching skimmed milk powder, both reconstituted in water. Participants will then undergo a series of tests to compare the effects of these two drinks on gastrointestinal fluid retention and motility as well as on gut comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Participants declare that they are of Chinese ethnicity as well as both of their biological parents
2. Women and men aged between 18 and 60 years
3. Body mass index (BMI ≥ 18.5 & <30 kg/m2)
4. Healthy: no medical conditions or previous gastrointestinal surgery which might affect study measurements (as declared by the participant)
5. Able to understand and to sign written informed consent prior to study entry
6. Informed consent signed
7. Meets all the criteria for MRI Scan
8. Can read and speak English

Exclusion Criteria:

1. Medically diagnosed milk allergy
2. Subjects not willing and/or not able to comply with scheduled visits and the requirements of the study protocol
3. Diagnosed with any gastrointestinal disorders
4. History of claustrophobia
5. Pregnant (defined by pregnancy test) or breast feeding
6. History or current psychiatric illness
7. History or current neurological condition (e.g. epilepsy)
8. Consumption of > 21 alcoholic drinks in a typical week (one serving is 0.4 dl of spirits, 1 dl of wine, or 3 dl of beer as declared by participant)
9. Currently smoking (as declared by participant)
10. Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance
11. Antibiotic use within the 4 weeks preceding the intervention
12. Probiotic & prebiotics use within the 2 weeks preceding the intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Small bowel water content | 0-315 minutes after investigational product (IP) or comparator product (CP) intake
  Small bowel water content measured via MRI and calculated using the trapezoidal rule (mL*min) at 45 minutes of interval
Gut motility | 0-315 minutes after IP or CP intake
  Maximum gut motility after product consumption (arbitrary unit) assessed via MRI performed every 45 min

SECONDARY OUTCOMES:
Gastric emptying | 0-315 minutes after IP or CP intake
  Time to empty half of the stomach contents (T1/2) (min) after product consumption assessed via MRI every 45 min
Retention rate of gastric content volumes | 0-315 minutes after IP or CP intake
  Retention rate (RR) of gastric content volumes (GCV) calculated as the percentage of GCV in the stomach at each time point relative to the GCV measured at time 0 (%) measured via MRI every 45 min
Oro-caecal transit | 0-315 minutes after IP or CP intake
  Time at appearance of a food bolus in the caecum (min) measured via MRI every 54 min
H2 levels | 0-315 minutes after IP or CP intake
  Time at which the level of breath H2 shows a sustained (3 consecutive measurements) rise > 20ppm over baseline after product consumption (min) measured every 22 min
Colonic volume | 0-315 minutes after IP or CP intake
  Colonic volume measured by MRI every 45 min after product consumption (mL*min)
Colonic gas production via MRI | 0-315 minutes after IP or CP intake
  Colonic gas measured by MRI every 45 min after product consumption (arbitrary unit)
Colonic gas production via breath test | 0-315 minutes after IP or CP intake
  Breath gas measurements (H2 and CH4) measured every 45 min after product consumption (ppm*min)
Colonic water content | 0-315 minutes after IP or CP intake
  Colonic water content measured via MRI every 45 minutes after product consumption (mL*min)
T1 relaxation time | 0-315 minutes after IP or CP intake
  T1 relaxation time of ascending colon measured measured every 45 min via MRI after product consumption (ms)
Bristol stool | 3 days before and after after IP or CP intake
  Bowel movements & stool consistency measured using a Bristol stool diary
GI symptoms | 0-315 minutes after IP or CP intake
  Ordinal scoring of digestive symptoms rating via GI questionnaire composed of eight questions (score) administrated every 45 min after product consumption. Scores go from 0 to 3, 0 = not at all; 1 = mild (distinct but negligible); 2 = moderate (annoying); 3 = severe (disabling)

OTHER OUTCOMES:
Appetite | 0-315 minutes after IP or CP intake
  Appetite composite score calculated using answer to a VAS appetite questionnaire (4 questions) administrated every 45 min after product consumption. Scores go from 1 to 5, with higher scores meaning a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Irma Silva Zolezzi, Study Director — Societé des Produits Nestlé SA
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No